CLINICAL TRIAL: NCT00907114
Title: Efficacy and Safety of Topic Ketorolac to Treat Center Point Thickness Secondary to Panphotocoagulation in Proliferative Diabetic Retinopathy
Brief Title: Topic Ketorolac Added to Panphotocoagulation in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Virgilio Lima Gomez, PhD, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HJM 1667/09.03.24
Record Dates: First submitted 2009-05-19; First posted 2009-05-22 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Proliferative Diabetic Retinopathy; Macular Edema
Keywords: proliferative diabetic retinopathy; macular edema; panphotocoagulation; topic ketorolac; efficacy; treatment
MeSH Terms: conditions — Macular Edema | interventions — Ketorolac Tromethamine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac tromethamine (Active Comparator): ocular topic ketorolac used 4 times a day during a week after panphotocoagulation
  Interventions: Drug: Ketorolac tromethamine
- Polivynilic alcohol (Placebo Comparator): ocular lubricant drops 4 times a day during one week after panphotocoagulation
  Interventions: Drug: Polivynilic alcohol

INTERVENTIONS:
Drug: Ketorolac tromethamine — Presentation 5 mg/ml; Dosage: one drop (0.25 mg) four times a day during one week after panphotocoagulation
  Other Names: Godek
  Arms: Ketorolac tromethamine
Drug: Polivynilic alcohol — Presentation: alcohol polivinilico 14 mg/ml; Dosage: one drop (0.7 mg alcohol polivinilico) four times a day during one week after panphotocoagulation
  Other Names: Acuafil
  Arms: Polivynilic alcohol

SUMMARY:
The purpose of this study is to determine the efficacy and safety of topic ketorolac in treatment for center point thickness secondary to panphotocoagulation in proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Panphotocoagulation is the standard treatment for proliferative diabetic retinopathy during 3 to 4 sessions within 2 weeks. This treatment reduces the incidence of severe visual loss in the long term. Nonetheless, it induces macular thickness that delays the conclusion of the treatment. This delay could coincide with vitreous hemorrhage which, in turn, may limit additional photocoagulation.

Topic ketorolac could limit the inflammatory reaction cause by panphotocoagulation and produce early benefits in the patient.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* proliferative diabetic retinopathy
* without macular edema
* adequate quality 6 mm fast macular map on the day of treatment
* visual capacity under subjective refraction before treatment
* signed of inform consent

Exclusion Criteria:

* ocular surgery in the last 4 months
* myopia over -6.00 diopters
* allergy to ketorolac or non-steroids antiinflammatory
* previous selective photocoagulation
* using non-steroids antiinflammatory or immunomodulators
* intraocular inflammatory
* any retinal disease different from diabetic retinopathy
* pregnancy
* actual corneal disease
* inadequate quality 6 mm fast macular map after the second visit
* inconsistency after the second visit
* adverse event of the drug
* remove of the inform consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
center subfield mean thickness using Stratus OCT measured in microns | baseline, 24, 48 and 168 hours after treatment

SECONDARY OUTCOMES:
center point thickness using Stratus OCT, measured in microns | baseline, 24, 48 and 168 hours after treatment
macular volume using Stratus OCT, measured in cubic millimeters | baseline, 24, 48 and 168 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Lima Gomez, MD, MSc, Study Chair — Hospital Juarez de Mexico; Dulce M Razo Blanco Hernandez, MD, Principal Investigator — Hospital Juarez de Mexico; Juan Asbun Bojalil, MD, PhD, Study Director — Hospital Juarez de Mexico
Locations (1):
- Virgilio Lima Gomez, Mexico City, Mexico City, Mexico